CLINICAL TRIAL: NCT01796548
Title: Extended-Release Oxybutynin in the Treatment of Neurogenic Detrusor Overactivity (RONDO)
Brief Title: Extended-Release Oxybutynin for the Treatment of Neurogenic Detrusor Overactivity
Acronym: RONDO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow rate of participant's enrollment
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015205; R016446OAB4011
Record Dates: First submitted 2013-01-30; First posted 2013-02-21 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-10

CONDITIONS: Detrusor Function, Overactive
Keywords: Detrusor function, overactive; Urinary incontinence; Oxybutynin; Lyrinel
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxybutynin Extended-Release (Experimental): Oxybutynin chloride 5, 10, 15 milligram (mg) per tablet 10-30 mg per day orally
  Interventions: Drug: Oxybutinin Extended-Release

INTERVENTIONS:
Drug: Oxybutinin Extended-Release — Oxybutynin chloride 5, 10, 15 milligram (mg) per tablet 10-30 mg per day orally
  Other Names: Lyrinel

SUMMARY:
The purpose of this study is to evaluate the effects and tolerability (how well a participant can stand a particular medicine or treatment) of flexible dose Oxybutynin Extended-Release (OXY-ER, Lyrinel) including safety and quality of life assessment in participants with neurogenic detrusor overactivity (NDO - the nerves mediating the detrusor muscle do not work properly leading to frequent feeling of need to urinate during the day, night, or both).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single arm, prospective (study following participants forward in time), multi-center study of participants with NDO. The initial dose of Oxybutynin ER will be 10 milligram (mg) and will be titrated to a maximum of 30 mg. Dosage will be adjusted in 5-mg increments at approximately 14-day intervals until continence is achieved or the participant cannot tolerate side effects. The duration of participation in the study will be 12 weeks. The study will consist of 6 visits: baseline, Weeks 2, 4, 6, 8 and 12. Week 4 and Week 8 will be telephone visits. Overall safety and efficacy of Oxybutinin ER will be assessed as well as safety and efficacy during the titration and maintenance phases. The efficacy of treatment will be assessed using urodynamic parameters (the force and flow of urine) and clinical parameters (voiding diary and catheterization [use or insertion of a tubular device to drain the bladder] schedules). The quality of life will also be monitored in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overactive bladder as a result of neurogenic condition, for example following spinal cord injury, multiple sclerosis (slowly worsening disorder of the central nervous system that causes symptoms such as weakness, incoordination, numbness, problems talking and problems seeing), Parkinson's disease (a progressive disorder of the central nervous system, seen usually in older persons, in which there is slow movement [due to muscle weakness], trembling and sweating), or cerebrovascular accidents (CVAs - stroke-sudden loss of blood supply to brain)
* Women must not be pregnant and be of either non-childbearing potential or is using adequate means of birth control
* Overactive bladder symptoms and/or has urge incontinence episodes
* Must have normal results on urine culture tests and on urinalysis
* ECOG (Eastern Cooperative Oncology Group) performance status score of less than or equal to 3

Exclusion Criteria:

* Participants with 1 or more treatable or conditions, other than neurogenic bladder dysfunction, that may cause urinary incontinence or urgency
* Any medical or unstable condition that precludes their participation in the study or may confound the outcome of the study (participants with or at risk for urinary retention, gastric retention or uncontrolled narrow angle; heart failure or kidney failure; diabetes mellitus; abnormal muscle weakness [myasthenia gravis]; paralysis or inactivity in the intestines that prevents material moving through the gut [intestinal atony or paralytic ileus]; severe inflammation of the bowel [ulcerative colitis] sudden expansion of the large intestine seen in advanced ulcerative colitis or Crohn's disease [toxic megacolon]; history of major lower urinary tract surgery [transurethral resection will be excluded])
* Hypersensitivity to the investigational drug or any of its ingredients (eg, lactose)
* Pregnant or breast feeding female
* Significant bacteriuria (presence of bacteria in the urine) or pyuria (presence of white blood cells) in the urine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (3):
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Phathumwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxybutynin: Participants received an initial dose of extended release (ER) oxybutynin chloride 10 milligram (mg) orally once daily, with an increment of 5 mg in the dosage, at an approximate 14-days interval to a maximum of 30 mg per day, until continence was achieved for the last 2 days of interval. Dose was decreased by 5 mg if there were intolerable side effects. The participants then continued the maintenance dose to 12-week treatment.
Period: Overall Study
Arm/Group | Oxybutynin
Started | 17
Treated | 15
Completed | 14
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- Oxybutynin: Participants received an initial dose of extended release (ER) oxybutynin chloride 10 milligram (mg) orally once daily, with an increment of 5 mg in the dosage, at an approximate 14-days interval to a maximum of 30 mg per day, until continence was achieved for the last 2 days of interval. Dose was decreased by 5 mg if there were intolerable side effects. The participants then continued the maintenance dose to 12-week treatment. 'Number of participants analyzed for the baseline characteristic was intent-to-treat (ITT) population which included all randomly assigned participants who received at least 1 dose of study medication and fulfilled all eligibility criteria.'
Arm/Group | Oxybutynin
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Maximal Detrusor Pressure [Mean (Standard Deviation); unit: Centimeter of water] — Maximal detrusor pressure represents the maximum pressure (peak amplitude) in the bladder during the first involuntary contraction of the bladder muscle. Detrusor pressure is the component of intravesical (in the bladder) pressure that is created by forces in the bladder wall (passive and active). It was estimated by subtracting abdominal pressure from intravesical pressure.
  Centimeter of water | 57.7 (28.1)

OUTCOME MEASURES:

1. Primary Outcome: Maximal Detrusor Pressure
Description: Maximal detrusor pressure represents the maximum pressure (peak amplitude) in the bladder during the first involuntary contraction of the bladder muscle. Detrusor pressure is the component of intravesical (in the bladder) pressure that is created by forces in the bladder wall (passive and active). It was estimated by subtracting abdominal pressure from intravesical pressure.
Time Frame: Week 12
Population: The Intent-to treat (ITT) population included all randomly assigned participants who received at least 1 dose of study medication and fulfilled all eligibility criteria.
Measure: Mean (Standard Deviation); unit: Centimeter of water
Arm/Group | Oxybutynin
Number analyzed (Participants) | 15
Centimeter of water | 42.8 (29.7)

2. Secondary Outcome: Maximal Cystometric Capacity (MCC)
Description: MCC represents the maximum volume of urine the bladder holds.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Milliliter (ml)
Arm/Group | Oxybutynin
Number analyzed (Participants) | 15
Milliliter (ml)
  Baseline | 169.9 (55.2)
  Week 12 | 268.8 (150.6)

3. Secondary Outcome: Detrusor Leakpoint Pressure
Description: Detrusor leakpoint pressure is the level of pressure at which leakage of urine through the urethra occurs as the bladder fills without an increase in abdominal pressure. This was a measure of both strength of the urethral sphincters and compliance of the detrusor muscle.
Time Frame: Baseline and Week 12
Population: Data for this outcome measure is not reported because the data was not collected and included in Case Report Form (CRF).
Arm/Group | Oxybutynin
Number analyzed (Participants) | 0

4. Secondary Outcome: Post-Void Residual Urine Volume
Description: Post-void residual urine volume is the amount of urine remaining in the bladder after void completion.
Time Frame: Baseline and Week 12
Population: ITT population. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for this measure at a particular time point.
Measure: Mean (Standard Error); unit: Milliliter (ml)
Arm/Group | Oxybutynin
Number analyzed (Participants) | 7
Milliliter (ml)
  Baseline (n= 7) | 112.1 (79.8)
  Week 12 (n= 4) | 184.5 (108.1)

5. Secondary Outcome: Reflex Volume
Description: Reflex volume is the infused volume that induces the first detrusor contraction.
Time Frame: Baseline and Week 12
Population: Data for this outcome measure is not reported because the data was not collected and included in Case Report Form (CRF).
Arm/Group | Oxybutynin
Number analyzed (Participants) | 0

6. Secondary Outcome: Urge Incontinence Episodes
Description: Urge incontinence episodes were reported. Urge urinary incontinence is the complaint of involuntary leakage accompanied by or immediately preceded by urgency with sudden feeling to go to toilet.
Time Frame: Baseline, Week 4 and Week 12
Population: ITT population. Here "n" signifies participants who were evaluable for this measure at a particular time point.
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Oxybutynin
Number analyzed (Participants) | 14
Episodes
  Baseline (n=14) | 8.8 (11.0)
  Week 4 (n=13) | 5.0 (11.4)
  Week 12 (n=13) | 4.9 (11.9)

7. Secondary Outcome: Total Incontinence Episodes
Description: Episodes of total urinary incontinence were reported. Urinary incontinence is the complaint of any involuntary leakage of urine.
Time Frame: Baseline, Week 4 and Week 12
Population: ITT population. Here "n" signifies participants who were evaluable for this measure at a particular time point. This study is early terminated and there were some missing data for total incontinence which lead to decrease value of total incontinence.
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Oxybutynin
Number analyzed (Participants) | 14
Episodes
  Baseline (n=14) | 7.4 (10.7)
  Week 4 (n=13) | 4.2 (11.5)
  Week 12 (n=13) | 4.8 (12.0)

8. Secondary Outcome: Percentage of Participants With no Episodes of Urge-Urinary Incontinence
Description: Percentage of participants with no episodes of urge urinary incontinence was reported. Urge urinary incontinence is the complaint of involuntary leakage accompanied by or immediately preceded by urgency.
Time Frame: Baseline, Week 4 and Week 12
Population: Data was not reported for this OM, as data was not analyzed because of change in the planned analysis of the study.
Arm/Group | Oxybutynin
Number analyzed (Participants) | 0

9. Secondary Outcome: King Health Questionnaire Score
Description: King Health Questionnaire assesses the physical and psycho-social aspects of the disease state. It is a self-administered questionnaire containing 21 questions scored in 9 domains (general health perception, incontinence impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep or energy, and severity of urinary symptoms). All domains were assessed in a range: 0-100, where 0=best outcome/response and 100=worst outcome or response. Lower scores indicates better outcome or response.
Time Frame: Baseline and Week 12
Population: ITT population. Here "N" signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxybutynin
Number analyzed (Participants) | 14
Units on a scale
  Baseline: General Health Perceptions | 53.5 (21.6)
  Baseline: Impact of Life | 76.1 (30.5)
  Baseline: Role Limitations | 66.7 (36.4)
  Baseline: Physical Limitations | 73.8 (22.4)
  Baseline: Social Limitations | 58.7 (29.0)
  Baseline: Personal Relationships | 66.7 (35.6)
  Baseline: Emotions | 57.1 (36.1)
  Baseline: Sleep or Energy | 51.2 (24.9)
  Baseline: Incontinence Severity | 44.0 (31.3)
  Week 12: General Health Perceptions | 35.7 (16.2)
  Week 12: Impact of Life | 59.5 (29.8)
  Week 12: Role Limitations | 63.1 (34.7)
  Week 12: Physical Limitations | 66.7 (27.7)
  Week 12: Social Limitations | 60.7 (32.5)
  Week 12: Personal Relationships | 30.9 (33.9)
  Week 12: Emotions | 41.3 (29.7)
  Week 12: Sleep or Energy | 42.9 (33.1)
  Week 12: Incontinence Severity | 33.9 (26.0)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Arm/Group | Oxybutynin
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxybutynin (N=15)
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxybutynin (N=15)
Pollakiuria (Renal and urinary disorders) | 1
Dry mouth (Gastrointestinal disorders) | 11
Urinary tract infection (Infections and infestations) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Vomitting (Gastrointestinal disorders) | 1
Nerve compression (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have first to present the data of Clinical Trial (CT) without approval from the Institution or PI. If the Institution and PI wish to publish data from CT, a copy of the same must be provided to Sponsor for review at least 60 days prior to submission. No paper with Confidential Information will be submitted with Sponsor's prior written consent. If requested in writing, Institution and PI will withhold publication for up to an additional 60 days to allow filing of patent application.